CLINICAL TRIAL: NCT01844063
Title: Clinical Comparison of Safety and Efficacy of Allogeneic Umbilical-Cord and Bone Marrow-derived Mesenchymal Stem Cells Transplantation for HBV-related Liver Failure
Brief Title: Safety and Efficacy of Diverse Mesenchymal Stem Cells Transplantation for Liver Failure
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Qi Zhang, MD, Deputy Director, Office of International Cooperation & Exchange Office of Hongkong, Macao & Taiwan Affairs, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: The Third Affiliated Hospital
Record Dates: First submitted 2013-04-20; First posted 2013-05-01 (Estimated); Last update posted 2013-07-08 (Estimated); Status verified 2013-07

CONDITIONS: Liver Failure
MeSH Terms: conditions — Liver Failure | interventions — Congresses as Topic; Antiviral Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Conventional treatment (Experimental): Participants will receive conventional treatment and then be followed until the week 72 study visit.
  Interventions: Drug: Conventional treatment
- Conventional plus BM-MSC treatment (Experimental): Participants will receive conventional treatment plus a dose of BM-MSC(each subgroups with a different dose ) and then be followed until the week 72 study visit.
  Interventions: Genetic: Conventional plus BM-MSC treatment
- Conventional plus UC-MSC treatment (Experimental): Participants will receive conventional treatment plus a dose of UC-MSC(each subgroups with a different dose ) and then be followed until the week 72 study visit.
  Interventions: Genetic: Conventional plus UC-MSC treatment

INTERVENTIONS:
Genetic: Conventional plus BM-MSC treatment — Received conventional treatment and bone marrow mesenchymal stem cells transplantation by peripheral vein slowly for 30minutes. (1×10e5/Kg,1×10e6/Kg,or 1×10e7/Kg, once a week, 8 times).
  Arms: Conventional plus BM-MSC treatment
Genetic: Conventional plus UC-MSC treatment — Received conventional treatment and bone marrow mesenchymal stem cells transplantation by peripheral vein slowly for 30minutes. (1×10e5/Kg,1×10e6/Kg,or 1×10e7/Kg, once a week, 8 times)
  Arms: Conventional plus UC-MSC treatment
Drug: Conventional treatment — Received conventional treatment including:
  A.antiviral drugs(Entecavir,Lamivudine,Adefovir dipivoxil,et al); B.Hepatoprotective drugs(Ademetionine1,4-butanethiosulfonate for Injection, Reduced Glutathione for Injection,Polyene Phosphatidylcholine, et al); C.Plasma.
  Other Names: Antiviral drugs; Hepatoprotective drugs; Plasma
  Arms: Conventional treatment

SUMMARY:
HBV-related liver failure (HBV-LF), a dramatic clinical syndrome, is characterized with massive necrosis of liver cells. Liver transplantation might be the most effective therapy for HBV-LF. However, there are a lot of problems such as lack of donors, surgical complications, transplant rejection, and high cost, which could limit the application of liver transplantation. It is demonstrated that mesenchymal stem cells could directionally differentiate into hepatocytes and cholangiocytes in injured liver, as well as reduce inflammation of the liver by immune regulation. In this study, we assess the safety and efficacy of human bone marrow and umbilical cord mesenchymal stem cells transplantation for patients with HBV-LF.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years
* Liver failure
* Negative pregnancy test (female patients in fertile age)
* Written consent
* HBsAg positive
* TB≥171 μmol/L or ascend ≥17.1 μmol/L/per day,
* INR≥1.5 or 20%<PTA≤40%
* 17≤MELD score≤30

Exclusion Criteria:

* Hepatocellular carcinoma or other malignancies
* Severe problems in other vital organs(e.g.the heart,renal or lungs)
* Pregnant or lactating women
* Severe bacteria infection
* Anticipated with difficulty of follow-up observation
* Liver failure caused by other reasons, such as autoimmune diseases, alcohol, drug and so on
* Other candidates who are judged to be not applicable to this study by doctors

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2013-07; Primary Completion 2016-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
survival rate | 72 weeks
  The survival rate and time

SECONDARY OUTCOMES:
Liver function | 72 weeks after treatment
  The levels of serum Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST),Cholinesterase (CHE) ,Total Bilirubin(TB),Direct Bilirubin(DB), Serum Albumin （ALB）
Marker of liver cancer | 72 weeks after treatment
  The level of alpha-fetoprotein (AFP)
The degree of hepatic necrosis | 2 years after treatment
  The levels of Prothrombin Activity (PA) and Prothrombin Time (PT)
The improvement of symptoms | 72 weeks after treatment
  The improvement of clinical symptoms [including appetite, debilitation, abdominal distension, edema of lower limbs, et al
The score for Model for End-Stage Liver Disease | 72 weeks after treatment
The improvement of immune function | 72 weeks after treatment
  cluster of differentiation 4 (CD4+)T/ cluster of differentiation 8 (CD8+)T,T helper cell 1 (Th1)/ T helper cell 1(Th2),natural killer cell(NK),natural killer T(NK T),interleukin-1β(IL-1β),interleukin-4(IL-4),interleukin-6(IL-6),interleukin-8(IL-8),interleukin-12(IL-12),interleukin-15(IL-15),interleukin-17A(IL-17A),Tumor necrosis factor-alpha (TNF-α),Interferon-gamma (IFN-γ)
complications | Between 0 to 8 hours after MSC transfusion
  The occurrence of complications [including body temperature, tetter and allergy]
The incidence of hepatocellular carcinoma | 72 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qi Zhang, Doctor, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Qi Zhang, Guangzhou, Guangdong, China